CLINICAL TRIAL: NCT04505592
Title: Tenecteplase With Concomitant Anticoagulation for Severe Acute Respiratory Failure in Patients With COVID-19
Brief Title: Tenecteplase in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hooman Poor (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Hooman Poor, Assistant Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 20-1764
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Results first posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; Respiratory Failure; ARDS
Keywords: COVID-19; ARDS; thrombolysis; tenecteplase
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Tenecteplase

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 ratio to treatment or control in blocks of 15, performed twice per dose (low and high) with randomization stratified by site.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and study investigators will be blinded to subject treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenecteplase (Experimental): First 20 patients randomized to treatment will receive tenecteplase 0.25 mg/kg (maximum 25 mg). Last 20 patients randomized to treatment will receive tenecteplase 0.50 mg/kg (maximum 40 mg).
  Interventions: Drug: Tenecteplase
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenecteplase — First 20 patients randomized to treatment arm will receive 0.25 mg/kg of tenecteplase. Next 20 patients randomized to treatment arm will receive 0.50 mg/kg of tenecteplase. Both will receive concomitant heparin to maintain activated partial thromboplastin time between 2.0 and 2.5 upper limit of normal.
  Arms: Tenecteplase
Drug: Placebo — Patients will receive placebo with concomitant heparin to maintain activated partial thromboplastin time between 2.0 and 2.5 upper limit of normal.
  Arms: Placebo

SUMMARY:
This is a placebo-controlled, double blind, randomized, Phase II dose escalation study intended to evaluate the potential safety and efficacy of tenecteplase for the treatment of COVID-19 associated respiratory failure. The hypothesis is that administration of the drug, in conjunction with heparin anticoagulation, will improve patients' clinical outcomes.

DETAILED DESCRIPTION:
Patients with COVID-19 who suffer from acute hypoxemic respiratory failure have a poor prognosis. COVID-19 has been associated with a hyperinflammatory and hypercoagulable state, leading to a range of thromboembolic complications from pulmonary embolism to ischemic stroke. Furthermore, emerging data suggest that the associated acute respiratory failure is, at least in part, due to pulmonary vascular disease caused by micro- and/or macro-emboli, creating pulmonary vascular shunting and dead-space ventilation. In this placebo-controlled, double blind, randomized, Phase II dose escalation study, we plan to evaluate the clinical efficacy and safety of low-dose IV bolus tenecteplase together with anticoagulation compared with control patients on therapeutic anticoagulation alone in hospitalized adults diagnosed with COVID-19 respiratory failure with elevated D-dimer. We believe these patients can be successfully treated without significantly increasing the risk of major bleeding while improving recovery rates, shorten hospitalization time, and perhaps ultimately prove to improve survival.

ELIGIBILITY:
Inclusion Criteria

* Patient/legally authorized representative has completed the Informed Consent Form
* Age ≥18 years
* Ability to comply with the study protocol, in the investigator's judgment
* Respiratory failure secondary to COVID-19 requiring mechanical ventilation for no greater than 24 hours, or high-flow nasal cannula (HFNC),non-rebreather (NRB) mask or non-invasive positive pressure ventilation (NIPPV) for no greater than 48 hours
* Confirmed infection with SARS-CoV-2 virus (PCR positive within 14 days)
* Elevated D-dimer (>6 times upper limit of normal within past 72 hours)
* For patient who are intubated >12 hours prior to randomization or with any evidence of neurologic deficit a head CT within 12 hours demonstrating no evidence of acute or subacute infarct or hemorrhage

Exclusion Criteria

* Current participation in another investigational drug study within the prior 7 days
* Known hypersensitivity or allergy to any ingredients of tenecteplase
* Active internal bleeding
* Known bleeding diathesis
* Use of one of the new oral anticoagulants within the last 48 hours (dabigatran, rivaroxaban, apixaban, edoxaban)
* Treatment with a thrombolytic within the last 3 months prior to randomization (exception for the use of Cathflo alteplase for occlusions of central venous catheters)
* Baseline platelet count <80,000/L (results must be available prior to treatment)
* Baseline blood glucose >400 mg/dL (22.20 mmol/L)
* Baseline blood glucose <50 mg/dL needs to be normalized prior to randomization
* Intracranial or intraspinal surgery or trauma within 2 months
* Other, non-COVID-19 related, serious, advanced, or terminal illness (investigator judgment) or life expectancy is less than 6 months
* History of acute ischemic stroke in the last 90 days
* History of intracranial bleeding, including hemorrhagic stroke
* Presumed septic embolus; suspicion of bacterial endocarditis
* Mechanical ventilation > 24 hours, HFNC, NRB, NIPPV, or any combination, for greater than 48 hours
* Mechanical ventilation, HFNC, NRB, or NIPVV (for reasons other than obstructive sleep apnea) within the prior 30 days (excluding 48 hours prior to randomization)
* Moribund status suggesting imminent vascular collapse and inability to survive > 72 hours (investigator determination)
* Uncontrolled hypertension defined as systolic BP > 180 mm Hg and/or diastolic BP > 110 mm Hgb
* Age > 75 years
* History of traumatic brain injury within 2 months
* Recent head trauma with fracture or brain injury
* History of Heparin Induced Thrombocytopenia (HIT) and/or other hereditary or acquired hemorrhagic diathesis or coagulation factor deficiency
* INR > 2 or recent oral anticoagulant therapy with INR >1.7
* Pregnancy or lactation within the prior 30 days; women of childbearing age (<55 years old) should have documentation of a negative pregnancy test
* Chronic liver disease defined as > Childs-Pugh Class B
* Atrial fibrillation, mitral stenosis, or known left heart thrombosis
* Any other condition that, in the opinion of the investigator, precludes administration of tenecteplase or poses a significant hazard to the patient receives tenecteplase

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Poor, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; J Mocco, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in a tertiary academic hospital in New York City.
Groups:
- Tenecteplase: Tenecteplase 0.25 mg/kg (maximum dose of 25 mg) And received concomitant heparin to maintain activated partial thromboplastin time between 2.0 and 2.5 upper limit of normal.
- Placebo: Patients received placebo with concomitant heparin to maintain activated partial thromboplastin time between 2.0 and 2.5 upper limit of normal.
Period: Overall Study
Arm/Group | Tenecteplase | Placebo
Started | 8 | 5
Completed | 6 | 4
Not Completed | 2 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenecteplase | Placebo | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.5 [55 to 71] | 71 [52 to 73] | 69 [52 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 3 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 35 [31 to 39] | 26 [24 to 27] | 31 [26 to 37]
Hypertension [Count of Participants; unit: Participants] | 6 | 3 | 9
Diabetes [Count of Participants; unit: Participants] | 2 | 1 | 3
Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 3 | 0 | 3
Obstructive Sleep Apnea [Count of Participants; unit: Participants] | 1 | 0 | 1
Respiratory Support [Count of Participants; unit: Participants] — Participants can have more than 1 type of respiratory support at baseline
  Participants
    Mechanical ventilation | 1 | 0 | 1
    high-flow nasal cannula (HFNC) | 4 | 3 | 7
    non-rebreather (NRB) | 1 | 0 | 1
    non-invasive positive pressure ventilation (NIPPV) | 2 | 3 | 5
Steroids [Count of Participants; unit: Participants] | 8 | 5 | 13
Remdesivir [Count of Participants; unit: Participants] | 7 | 2 | 9
P/F Ratio [Median (Inter-Quartile Range); unit: Ratio] — Ratio of arterial pO2 over fraction of inspired oxygen that the patient is receiving. Normal P/F Ratio is ≥ 400.
  300 to 200 is considered mild ARDS
  200 to 100 is considered moderate ARDS
  Anything below 100 is considered severe ARDS.
  Ratio | 80 [67 to 111] | 87 [72 to 131] | 83 [68 to 119]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free of Respiratory Failure
Description: The number of patients free of respiratory failure defined as not requiring high flow nasal cannula, non-rebreather, noninvasive positive pressure ventilation, or mechanical ventilation at 28 days
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 5 | 2

2. Primary Outcome: Number of Participants With Occurrences of Bleeding
Description: Safety as assessed by number of participants with occurrences of intracranial bleeding or major bleeding
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 2 | 1

3. Secondary Outcome: Number of Participants With In-hospital Deaths at 14 Days
Description: Number of patients who expired in the hospital within the first 14 days of their participation in the study
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 2 | 1

4. Secondary Outcome: Number of Participants With Death at 28 Days
Description: Number of participants who expired by 28 days/end of study
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 2 | 1

5. Secondary Outcome: Number of Ventilator-free Days
Description: Number of ventilator-free days in 28 days period
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
days | 18 [3 to 28] | 19 [9 to 28]

6. Secondary Outcome: Number of Respiratory Failure-free Days
Description: Respiratory failure-free defined as not requiring high flow nasal cannula, non-rebreather, noninvasive positive pressure ventilation, or mechanical ventilation. Number of respiratory failure-free days in 28 days period.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
days | 0.5 [0 to 3] | 3 [1 to 5]

7. Secondary Outcome: Number of Vasopressor-free Days
Description: Number of vasopressor-free days over 28 days period
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
days | 9 [4.6 to 18.5] | 9 [9 to 18]

8. Secondary Outcome: Number of Vasopressor Doses at 24 Hours
Time Frame: 24 hours and 72 hours
Measure: Number; unit: doses
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
doses
  24 hours | 0 | 0
  72 hours | 0 | 0

9. Secondary Outcome: P/F Ratio
Description: The P/F ratio equals the arterial pO2 ("P") from the ABG divided by the FIO2 ("F") - the fraction (percent) of inspired oxygen that the patient is receiving expressed as a decimal (40% oxygen = FIO2 of 0.40).
  Ratio of arterial pO2 over fraction of inspired oxygen that the person is receiving.
  Normal P/F Ratio is ≥ 400.
  300 to 200 is considered mild ARDS
  200 to 100 is considered moderate ARDS
  Anything below 100 is considered severe ARDS.
Time Frame: 24 hours and 72 hours
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
Ratio
  24 hours | 89 [68 to 92] | 97 [89 to 146]
  72 hours | 89 [63 to 91] | 78 [77 to 137]

10. Secondary Outcome: Number of ICU-free Days
Description: Number of days the patient spent outside the ICU
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
days | 1 [1 to 7] | 1 [1 to 5]

11. Secondary Outcome: Hospital Length of Stay
Description: Length of time the patient spent in the hospital, including ICU
Time Frame: up to 29 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
days | 11 [7.8 to 29] | 13 [12 to 29]

12. Secondary Outcome: Number of Participants With New-onset Renal Failure
Description: Number of patients who experienced renal failure during the course of the study
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 0 | 3

13. Secondary Outcome: Number of Participants With Need for Renal Replacement Therapy
Description: Number of patients who underwent renal replacement treatment for their renal failure
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 8 | 5
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Tenecteplase | Placebo
All-Cause Mortality (participants affected / at risk) | 2/8 | 1/5
Serious Adverse Events (participants affected / at risk) | 4/8 | 4/5
Other Adverse Events (participants affected / at risk) | 3/8 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=8) | Placebo (N=5)
Cardiogenic shock (Cardiac disorders) | 1 | 0
ST Elevation Myocardial Infarction (STEMI) (Cardiac disorders) | 1 | 0
Worsening respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Large retroperitoneal hematoma with hgb drop (Blood and lymphatic system disorders) | 1 | 0
Intubation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhagic shock (Blood and lymphatic system disorders) | 0 | 1
Death (General disorders) | 1 | 1
Compartment syndrome (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=8) | Placebo (N=5)
Renal failure (Renal and urinary disorders) | 1 | 1
Decreased hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Mild oral bleeding (Blood and lymphatic system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Bleeding from mouth and wrist (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT04505592/Prot_SAP_000.pdf